CLINICAL TRIAL: NCT01312142
Title: Changes of Weaning Parameter in Weaning Failure Patient After Tracheostomy as a Predictor of Subsequent Weaning
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201012007RC
Record Dates: First submitted 2011-03-08; First posted 2011-03-10 (Estimated); Last update posted 2011-12-20 (Estimated); Status verified 2011-12

CONDITIONS: Weaning Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- patients with difficult weaning

SUMMARY:
Weaning from mechanical ventilator is an essential element in the care of critically ill intubated patients receiving mechanical ventilation. It covers the entire process of liberating the patient from mechanical support and from endotracheal tube.

The process of weaning involves two-step strategies: 1. Assessment of readiness for weaning, including physiological measurement, such as maximum inspiratory pressure, tidal volume, respiratory rate and etc. 2. Spontaneous breathing trial.

Tracheostomy has become an increasingly common intervention in ICUs, especially for patients with prolonged mechanical ventilator support.

Tracheostomy may reduce work of breathing by improving some aspects of pulmonary mechanics, such as reducing dead space and decreasing airway resistance, but to date, there is no evidence that this is linked to reduction in weaning time or length of stay.

The investigators believe such improvement in pulmonary mechanic, which may reflect in the weaning parameter that respiratory therapist measured before weaning program, may be different from that measured before tracheostomy creation.

The investigators therefore hypothesized that the improvement in pulmonary mechanic for patients with weaning failure after tracheostomy may reflect on weaning parameters, and that this improvement may be able to predict the subsequent successful weaning from mechanical ventilator support.

Hereby the investigators perform a prospective single-center study to investigate the changes of weaning parameters in difficult weaning patients after tracheostomy as a predictor of subsequent successful weaning.

DETAILED DESCRIPTION:
Weaning from mechanical ventilator is an essential element in the care of critically ill intubated patients receiving mechanical ventilation. It covers the entire process of liberating the patient from mechanical support and from endotracheal tube1. The process of weaning involves two-step strategies: 1. Assessment of readiness for weaning, including physiological measurement, such as maximum inspiratory pressure, tidal volume, respiratory rate and etc. 2. Spontaneous breathing trial. The incidence of successful weaning is estimated around 68.8%.

Despite there is no consensus on the optimal timing of tracheostomy, patients with prolonged trans-laryngeal intubation are finally succumbed to tracheostomy, as prolonged trans-laryngeal intubation causes tissue trauma, promotes bacterial translocation and infection, making tracheostomy an increasingly common intervention in ICUs. Meanwhile, tracheostomy may reduce work of breathing by improving some aspects of pulmonary mechanics, such as reducing dead space and decreasing airway resistance, but to date, there is no evidence that this is linked to reduction in weaning time or length of stay.

Ｗe believe such improvement in pulmonary mechanics, which may reflect in the weaning parameters that respiratory therapist measured before weaning program, may be different after tracheostomy creation, especially in those patient with weaning failure. Ｗe therefore hypothesized that there may be an improvement in pulmonary mechanic for patients with weaning failure after tracheostomy, and that this improvement may be able to predict the subsequent successful weaning from mechanical ventilator support. Hereby the investigators perform a prospective single-center study to investigate the changes of weaning parameters in weaning failure patients after tracheostomy as a predictor of successful weaning.

ELIGIBILITY:
Inclusion Criteria:

* All patients with prolonged mechanical ventilator support or difficult weaning who received tracheostomy subsequently.

Exclusion Criteria:

* Parturient
* Patient with upper airway obstruction
* Patients aged < 18 year old
* Patients who join other on going study

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with difficult weaning and received subsequent tracheostomy
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-04 (Estimated); Study Completion 2012-04 (Estimated)

PRIMARY OUTCOMES:
Changes of weaning parameters after tracheostomy | 5 days
  Weaning parameters are measured before and after tracheostomy creation too see if there is any changes

SECONDARY OUTCOMES:
To evaluate if changes in weaning parameters will predict successful weaning | 6 months
  We will first measure the changes of weaning parameters after tracheostomy. If changes do occur, we would like to evaluate if it will predict subsequent weaning feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: Jih-Shuin Jerng, MD, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Lim CK, Ruan SY, Lin FC, Wu CL, Chang HT, Jerng JS, Wu HD, Yu CJ. Effect of Tracheostomy on Weaning Parameters in Difficult-to-Wean Mechanically Ventilated Patients: A Prospective Observational Study. PLoS One. 2015 Sep 17;10(9):e0138294. doi: 10.1371/journal.pone.0138294. eCollection 2015. PMID 26379127